CLINICAL TRIAL: NCT04200534
Title: Improving the Quality of Smoking Cessation and Shared Decision Making for Lung Cancer Screening: A Cluster Randomized Trial
Brief Title: Centralized Lung Cancer EARly Detection Among Smokers (CLEAR Study)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0265; NCI-2019-05127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0265 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-19; First posted 2019-12-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-03

CONDITIONS: Smoking; Lung Cancer
Keywords: current smoker; health care provider; primary care doctor
MeSH Terms: conditions — Smoking; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (centralized care strategy) (Experimental): Participants receive counseling over the phone to help them quit smoking and learn about lung cancer screening over 15-20 minutes for 6-8 sessions over 8 weeks. Participants may also receive nicotine patches.
  Interventions: Drug: Nicotine Patch; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling
- Group II (usual care) (Active Comparator): Participants receive counseling on lung cancer screening and smoking cessation from primary care providers at health care visit.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care counseling
  Other Names: standard of care; standard therapy
  Arms: Group II (usual care)
Drug: Nicotine Patch — Given nicotine patches
  Other Names: NicoDerm CQ; Nicotine Skin Patch; Nicotine Transdermal Patch
  Arms: Group I (centralized care strategy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Tobacco Cessation Counseling — Receive counseling over the phone
  Arms: Group I (centralized care strategy)

SUMMARY:
This trial studies how well a centralized care strategy works in improving the quality of smoking cessation and shared decision making among patients who smoke and are considering lung cancer screening. The centralized care strategy is a model where smokers eligible for lung cancer screening are referred to a dedicated tobacco treatment program where they receive both the shared decision-making and initiate smoking cessation counseling prior to their visit with a primary care provider. Utilizing the centralized care model may work better in helping people quit smoking and make informed decisions about lung cancer screening compared to usual care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test the effectiveness of usual care (primary care providers with training in guideline-based smoking cessation and shared decision making) versus (vs.) centralized care (smoking cessation and shared decision making delivered remotely by trained counselors) on smoking abstinence and the quality of patients' decisions about lung cancer screening.

SECONDARY OBJECTIVES:

I. Evaluate the reach, acceptability, feasibility, and fidelity of the two smoking cessation and shared decision-making implementation models in meeting the requirements from Centers for Medicare & Medicaid Services (CMS) for the lung cancer screening patient counseling and shared decision making visit.

II. Conduct budget impact and cost-effectiveness analyses of the two implementation models for the smoking cessation and shared decision making to inform adoption of the intervention beyond the current study.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I (CENTRALIZED CARE): Participants receive counseling over the phone to help them quit smoking and learn about lung cancer screening over 15-20 minutes for 6-8 sessions over 8 weeks. Participants may also receive nicotine patches.

GROUP II (USUAL CARE): Participants receive counseling on lung cancer screening and smoking cessation from primary care providers at health care visit.

After completion of study, participants are followed up at 1, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Primary care patients
* PATIENTS: Upcoming primary care office visit
* PATIENTS: Current smoker
* PATIENTS: 30 plus (+) pack-year smoking history
* PATIENTS: English-speaking
* PROVIDERS: Primary health care providers
* PROVIDERS: Provide care to adults

Exclusion Criteria:

* PATIENTS: History of lung cancer by self-report

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence Questionnairre | Up to 12 weeks
  Participants achieving the primary abstinence endpoint at 12 weeks (higher 7-day point prevalence abstinence rates)
Lung Cancer Screening 12 items version | Up to 12 weeks
  Knowledge of lung cancer screening and benefits of smoking cessation

SECONDARY OUTCOMES:
Number of patients who received smoking cessation counseling and shared decision making over the number of patients consented to participate in the study | Up to 12 weeks
  Assessment of the reach of the intervention
Acceptability, appropriateness, and feasibility of the intervention measure (Weiner et al). | Up to 12 weeks
  Assessment of the feasibility of implementing the intervention
Fidelity checklist (11 items) | Up to 12 weeks
  Assessment of the feasibility of implementing the intervention
EuroQoL-5 dimensions | Up to 12 weeks
  Standardized measure of health-related quality of life used to generate patient utilities (will report lower decisional conflict, greater decision preparation, greater intention to stop smoking, and be more likely to make an attempt to stop smoking.)
Costs of implementing any smoking cessation plus shared decision making intervention | Up to 12 weeks
  Costs of personnel, hardware, and delivering materials to participants

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Volk, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas

REFERENCES:
- [Derived] Lowenstein LM, Shih YT, Minnix J, Lopez-Olivo MA, Maki KG, Kypriotakis G, Leal VB, Shete SS, Fox J, Nishi SP, Cinciripini PM, Volk RJ. A protocol for a cluster randomized trial of care delivery models to improve the quality of smoking cessation and shared decision making for lung cancer screening. Contemp Clin Trials. 2023 May;128:107141. doi: 10.1016/j.cct.2023.107141. Epub 2023 Mar 5. PMID 36878389
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04200534/ICF_000.pdf